CLINICAL TRIAL: NCT05123560
Title: First-trimester Preeclampsia Screening: Women's Perspectives
Brief Title: Women's Perspective on First-trimester Preeclampsia Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Cristina Trilla, Principal investigador, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-PRE-2021-23
Record Dates: First submitted 2021-10-08; First posted 2021-11-17 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Woman's Role; Preeclampsia; Screening
Keywords: Preeclampsia screening; First-trimester; Women's perception; Anxiety; Stress; Clinical practice
MeSH Terms: conditions — Pre-Eclampsia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women attending first-trimester ultrasound: All women attending their first-trimester ultrasound and meeting the inclusion criteria will be invited to participate
  Interventions: Other: Anonymous online questionnaire

INTERVENTIONS:
Other: Anonymous online questionnaire — A QR code qill be provided to access the online questionnaire

SUMMARY:
The aim of this study is to evaluate women's perception on first-trimester preeclampsia screening as it is performed currently in daily practice. Thus, the investigators will assess the degree of satisfaction regarding the information received previously to the date of screening, and on the same day the screening is performed (at the time of first-trimester scan).

Women's unsderstanding regarding preeclampsia screening will be evaluated by means of an anonymous online questionnaire. Anxiety and stress related to the results will also be assessed.

DETAILED DESCRIPTION:
Preeclampsia screening was established in Catalonia in 2018. However, little training for professionals (doctors and midwifes) was performed. Women's opinion regarding screening was not asked prior to its implementation, and most women no dot receive any information prior to be screened.

Women's opinion on their pregnancy follow-ups is important, but this aspect is often not included in clinical practice policies. Thus, the objective of the study is to evaluate women's perception regarding current clinical practice in screening of preeclampsia, and their degree of satisfaction.

Screening and risk-assessments during pregnancy are also a potential cause of stress for women. Anxiety and stress regarding preeclampsia screening results will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Older that 18 years old
* singleton pregnancy
* low risc of cromosomal abnormalities (<1/1100)
* normal first trimester ultrasound (no evidence of fetal malformations)

Exclusion Criteria:

- Pacients will diagnosed mental disorders (including depression and anxiaety disorder)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — this study is only for pregnant women, regardless of their gender perceived identity
Study Population: All pregnant women with a singleton pregnancy attending their first-trimester ultrasound and undergoing preeclampsia screening
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Perception on information prior to the appointment to screen | 11-14 weeks of pregnancy
  Number of Participants with a high satisfaction degree with the received information prior to screening assessed by Baker's questionnaire. Answers to Baker's questionnaire: 1) Strongly agree 2) Somewhat agree 3) Neither agree nor disagree 4) Somewhat disagree 5) Strongly disagree. None of the answers mean a better or worse outcome. The aim is to record and characterize women's perception.
Perception on information received the day of the screening | 11-14 weeks of pregnancy
  Number of Participants with a high satisfaction degree with the received information the day of the screening assessed by Baker's questionnaire. Answers to Baker's questionnaire: 1) Strongly agree 2) Somewhat agree 3) Neither agree nor disagree 4) Somewhat disagree 5) Strongly disagree. None of the answers mean a better or worse outcome. The aim is to record and characterize women's perception.

SECONDARY OUTCOMES:
Anxiety and stress related to the results of the preeclampsia screening | 11-14 weeks of pregnancy
  Number of Participants with high anxiety and stress levels after the screening assessed by short version of the State-Trait Anxiety Inventory (STAI). Answers to the STAI questionnaire: 1) Not at all 2) A little bit 3) Quite a bit 4) Extremely. Answers 1 and 2 suggest low stress levels and answers 3 and 4 suggest high stress levels. Final score to characterize stress levels will be obtained after considering all answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] O'Gorman N, Wright D, Poon LC, Rolnik DL, Syngelaki A, Wright A, Akolekar R, Cicero S, Janga D, Jani J, Molina FS, de Paco Matallana C, Papantoniou N, Persico N, Plasencia W, Singh M, Nicolaides KH. Accuracy of competing-risks model in screening for pre-eclampsia by maternal factors and biomarkers at 11-13 weeks' gestation. Ultrasound Obstet Gynecol. 2017 Jun;49(6):751-755. doi: 10.1002/uog.17399. Epub 2017 May 14. PMID 28067011
- [Background] Rolnik DL, O'Gorman N, Roberge S, Bujold E, Hyett J, Uzan S, Beaufils M, da Silva Costa F. Early screening and prevention of preterm pre-eclampsia with aspirin: time for clinical implementation. Ultrasound Obstet Gynecol. 2017 Nov;50(5):551-556. doi: 10.1002/uog.18899. No abstract available. PMID 28887883
- [Background] Simeone S, Lojo C, Garcia-Esteve L, Triunfo S, Crovetto F, Arranz A, Gratacos E, Figueras F. Psychological impact of first-trimester prevention for preeclampsia on anxiety. Prenat Diagn. 2015 Jan;35(1):60-4. doi: 10.1002/pd.4485. Epub 2014 Sep 22. PMID 25156501
- [Background] Luchian B, Neagu M, Luchian L, Vladareanu R. Preeclampsia screening from the patient's perspective. J Med Life. 2016 Jul-Sep;9(3):321-323. PMID 27974943
- [Background] Jorgensen JM, Hedley PL, Gjerris M, Christiansen M. Including ethical considerations in models for first-trimester screening for pre-eclampsia. Reprod Biomed Online. 2014 May;28(5):638-43. doi: 10.1016/j.rbmo.2014.01.013. Epub 2014 Feb 7. PMID 24631382
- [Background] Jorgensen JM, Hedley PL, Gjerris M, Christiansen M. Ethical issues related to screening for preeclampsia. Bioethics. 2014 Sep;28(7):360-7. doi: 10.1111/j.1467-8519.2012.02005.x. Epub 2012 Sep 20. PMID 22994561
- [Background] Baker R. Development of a questionnaire to assess patients' satisfaction with consultations in general practice. Br J Gen Pract. 1990 Dec;40(341):487-90. PMID 2282225
- [Background] Fernandez San Martin MI, Rebagliato Nadal O, de Gispert Uriach B, Roig Carrera H, Artigas Guix J, Bonay Valls B, Guix Font L, Turmo Tristan N. [Adaptation of a patient satisfaction questionnaire on medical and nursing care]. Aten Primaria. 2008 Dec;40(12):611-6. doi: 10.1016/s0212-6567(08)75694-4. Spanish. PMID 19100148
- [Background] Buela-Casal G, Guillen-Riquelme A. Short form of the Spanish adaptation of the State-Trait Anxiety Inventory. Int J Clin Health Psychol. 2017 Sep-Dec;17(3):261-268. doi: 10.1016/j.ijchp.2017.07.003. Epub 2017 Aug 14. PMID 30487901